CLINICAL TRIAL: NCT03351140
Title: Qualitative Interviews to Evaluate the PROMIS Physical Function Item Bank for Use in Oncology Clinical Trials
Brief Title: Patient-Reported Outcome Measurement Information System (PROMIS) Physical Function
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Health Research Associates, Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 207113
Record Dates: First submitted 2017-11-09; First posted 2017-11-22 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Neoplasms
Keywords: Multiple Myeloma; Patient-Reported Outcome Measurement Information System (PROMIS); Non-Small Cell Lung Cancer (NSCLC); Breast cancer; Diffuse Large B-Cell (DLBCL); Follicular Lymphoma; Prostate Cancer; Qualitative interview
MeSH Terms: conditions — Neoplasms; Multiple Myeloma; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Lymphoma, Follicular; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Subjects with breast cancer: Approximately 30 subjects who have confirmed diagnosis of breast cancer will be included in the study
  Interventions: Other: Qualitative Interviews; Other: PROMIS Physical Function Items
- Subjects with prostate cancer: Approximately 30 subjects who have confirmed diagnosis of prostate cancer will be included in the study
  Interventions: Other: Qualitative Interviews; Other: PROMIS Physical Function Items
- Subjects with NSCLC: Approximately 30 subjects who have confirmed diagnosis of NSCLC will be included in the study
  Interventions: Other: Qualitative Interviews; Other: PROMIS Physical Function Items
- Subjects with multiple myeloma: Approximately 30 subjects who have confirmed diagnosis of multiple myeloma excluding smoldering/asymptomatic multiple myeloma will be included in the study
  Interventions: Other: Qualitative Interviews; Other: PROMIS Physical Function Items
- Subjects with DLBCL or follicular lymphoma: Approximately 30 subjects who have confirmed diagnosis of DLBCL or follicular lymphoma will be included in the study
  Interventions: Other: Qualitative Interviews; Other: PROMIS Physical Function Items

INTERVENTIONS:
Other: Qualitative Interviews — Subjects will participate in a qualitative interview lasting up to 90 minutes. The interviews will include a concept elicitation component to explore details of the subject's perceived disease condition, functional limitations and impacts on daily life and health-related quality-of-life (HRQoL). In addition, a card sorting exercise will be used to evaluate the relevance and comprehension of PROMIS Physical Function items.
Other: PROMIS Physical Function Items — PROMIS Physical Function Items is a set of self-report measurement tools. The latest version of PROMIS Physical Function Items contains 165 items for self-assessment. PROMIS Physical Function Cancer Item Bank contains a subset of 45 items relevant to cancer subjects. Subjects will complete half of the PROMIS Physical Function Items during their enrollment visit and the other half of items prior to their interview.

SUMMARY:
The objective of this study is to conduct in-person qualitative interviews of subjects who have different tumor types to identify and assess relevant PROMIS physical function items that can be utilized in future studies. Health Research Associates (HRA) will conduct qualitative interviews in subjects with a variety of cancer types. PROMIS is a set of self-report measurement tools, developed by the United States (US) National Institutes for Health (NIH). The most recent version of PROMIS Physical Function Item Bank contains 165 items assessing a range of abilities and its subset, a 45-item PROMIS Function Cancer Item Bank which contains questions relevant to subjects with cancer. Approximately 150 subjects with five tumor types will be recruited. HRA will conduct the interviews that will be audio-recorded for transcription and analysis. Five tumor types that will be focused on are Breast, Prostate, Non-Small-Cell Lung Cancer (NSCLC), Multiple Myeloma, and Diffuse Large B-Cell (DLBCL) or Follicular Lymphoma. Interviews will be conducted in English language in private areas within clinic site or rented meeting facilities and will last approximately for 60-90 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a confirmed diagnosis of a primary tumor of one of the following: Breast Cancer, Prostate Cancer, NSCLC, Multiple Myeloma (excluding smoldering/asymptomatic multiple myeloma) and DLBCL or Follicular Lymphoma
* Subject is able to read, write, and speak English well enough to understand and complete Informed Consent Form (ICF) and take part in the interview process
* Subject has received treatment for their qualifying tumor within the prior 6 months, with the exception of treatment-naïve subjects who have been diagnosed within the past 6 months
* Subject is at least 18 years of age
* Subject has an estimated life expectancy of 3 months or greater

Exclusion Criteria:

* Subject has more than one current primary tumor
* Subject has a Stage 0 or in situ neoplasm
* Subject has known unstable and/or untreated brain metastasis
* Subject had major surgery within the last 30 days prior to enrolment that may be associated with changes in physical function. Open biopsy is considered a major surgery
* Subject has a current or past history of a personality disorder, bipolar disorder, schizophrenia or other psychotic disorder, obsessive compulsive disorder, cognitive disorder, post-traumatic stress disorder, or other mental deficit
* In the opinion of the site investigator or study director, subject has any medical condition or disorder that could compromise his/her ability to give written informed consent and/or prevent or interfere with the Subject's ability to successfully participate in a face-to-face interview and provide meaningful and non-confounded information about their experience with their qualifying tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with confirmed diagnosis of breast cancer or prostate cancer or NSCLC or multiple myeloma, DLBCL or Follicular Lymphoma will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2020-05-08 (Actual)

PRIMARY OUTCOMES:
Conduct qualitative patient interviews with a range of cancer patients across multiple tumor types to identify a subset of relevant PROMIS Physical Function items that can be utilized in future clinical trials | Approximately 90 minutes
  Number of interviews conducted. Demographic and clinical characteristics of subjects will include Eastern Cooperative Oncology Group (EGOC) status, current tumor status and latest line of treatment

SECONDARY OUTCOMES:
Number of subject expressions of a given concept | Approximately 90 minutes
  Evidence to support the content validity for the selected PROMIS Physical functional items will include the number of subject expressions of given concept.
Number of interviews to reach saturation of concept | Approximately 90 minutes
  Evidence to support content validity includes the number of interviews needed to reach saturation of concept, which is the point, after which no new relevant or important information emerges and collecting additional data will not add to the understanding of how patients perceive the concept of interest and the items in a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Mountlake Terrace, Washington, United States

IPD SHARING:
Plan to Share IPD: No